CLINICAL TRIAL: NCT05568485
Title: Biopsychosocial Exercise Model Via Telerehabilitation in Individuals With Rheumatic Disease During the COVID-19 Pandemic
Brief Title: Telerehabilitation in Individuals With Rheumatic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Sevim Öksüz, physiotherapist, Eastern Mediterranean University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO-18/1182
Record Dates: First submitted 2022-09-22; First posted 2022-10-05 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Rheumatic Diseases
Keywords: Biopsychosocial, rheumatology, remote care, holistic
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (Experimental): Telerehabilitation was applied to the group with rheumatism
  Interventions: Other: Telerehabilitation was applied to the group with rheumatism

INTERVENTIONS:
Other: Telerehabilitation was applied to the group with rheumatism — Telerehabilitation was applied to the group with rheumatism in 3 sessions a week for 24 weeks via a social texting program. The intervention sessions consisted of 10 minutes of dance therapy-authentic movement, 40 minutes of exercises, and 10 more minutes of dance therap

SUMMARY:
increasing the prevalence of exercise models designed in accordance with the biopsychosocial model is very important in terms of ensuring the sustainability of these models with telerehabilitation in periods such as epidemics and pandemics. The aim of this study was to investigate the effects of a biopsychosocial exercise model provided via telerehabilitation in individuals with rheumatic diseases during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Telerehabilitation was applied to the group with rheumatism in 3 sessions a week for 24 weeks via a social texting program. The intervention sessions consisted of 10 minutes of dance therapy-authentic movement, 40 minutes of exercises, and 10 more minutes of dance therapy. This exercise content was based on a biopsychosocial model, named the Cognitive Exercise Therapy Approach (BETY) which was used in the study, and it was a method that patients already practiced before the pandemic. At the beginning, at the 12th week and 24th week, the Health Assessment Questionnaire (HAQ), the Hospital Anxiety and Depression Scale (HADS), the BETY Biopsychosocial Questionnaire (BETY-BQ) were applied.

ELIGIBILITY:
Inclusion Criteria:

members of an exercise group before the pandemic at the physiotherapy and rehabilitation department of a university.

Exclusion Criteria:

* Individuals who had difficulty in cooperation

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
BETY Biopsychosocial Questionnaire (BETY-BQ | change will be assessed at 12th week and 24th week
  an assessment tool that evaluates biopsychosocial involvement and assesses pain, function, sexual behavior, and social and psychological aspects. The scoring of the questionnaire is made using a 5-point Likert system. Each item is scored as "0 = No, never, 1 = Yes, rarely, 2 = Yes, sometimes, 3 = Yes, often, or 4 = Yes, always". A high score indicates a low biopsychosocial status

SECONDARY OUTCOMES:
Health assessment questionnaire | change will be assessed at 12th week and 24th week
  It includes 20 questions and 8 components including dressing, sitting, eating, walking, hygiene, reaching out, comprehending, and activities of daily living. Each answer is rated between 0 and 3 points, "0 = No difficulty, 1 = Somewhat difficult, 2 = Very difficult, and 3 = I can never do it", and a high score indicates low functionality [18]. HAQ scores of >1 are considered to indicate the presence of disability
hospital qnxiety and depression scale | change will be assessed at 12th week and 24th week
  . It is a 14-item scale that consists of Anxiety (HADS-A) and Depression (HADS-D) subscales. The answer to each item is scored between 0 and 3 using the 4-point Likert scoring format, and each subscale has a score range between 0 and 21. Scores between 0 and 7 for each subscale are considered "normal", those between 8 and 10 are considered "mild anxiety/depression", and those from 11 to 21 are considered moderate-severe anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep İrem Bulut, MSc. Pt., Principal Investigator — Hasan Kalyoncu University; Nur Banu Karaca, MSc. Pt., Principal Investigator — Hacettepe University; Arzu Dağ, Principal Investigator — İstanbul Yeni Yüzyıl University; Yavuz Yakut, Prof.Dr., Study Director — Hasan Kalyoncu University; Sedat Kiraz, Prof. Dr., Study Director — Hacettepe University
Locations (1):
- Eastern Mediterranen University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No